CLINICAL TRIAL: NCT00858052
Title: Core Study of the Safety and Effectiveness of IDEAL IMPLANT(R) Saline-filled Breast Implants in Women Who Are Undergoing Primary Breast Augmentation or Replacement of Existing Augmentation Implants
Brief Title: Core Study of the Safety and Effectiveness of IDEAL IMPLANT(R) Saline-filled Breast Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ideal Implant Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G 080055
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Breast Implants
Keywords: breast implants; saline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- breast augmentation (Experimental): breast implant
  Interventions: Device: Saline-filled breast implant [IDEAL IMPLANT (R)]

INTERVENTIONS:
Device: Saline-filled breast implant [IDEAL IMPLANT (R)] — Breast augmentation
  Other Names: IDEAL IMPLANT (R) Saline-filled Breast Implant

SUMMARY:
The objective of this study is to determine the safety and effectiveness of the IDEAL IMPLANT in women who are undergoing primary breast augmentation or replacement of existing saline-filled or silicone gel-filled augmentation implants.

DETAILED DESCRIPTION:
For complete information about the clinical trial, see link in the reference section.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral primary breast augmentation-dissatisfaction with breast size
* Bilateral replacement augmentation-has had previous silicone saline-filled or gel-filled breast implants

Exclusion Criteria:

* Diagnosis of active cancer of any type
* Has ever been diagnosed with breast cancer
* Has pre-malignant breast disease
* Has tissue characteristics incompatible with an implant
* Has unrealistic or unreasonable expectations of the procedure results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Determine the safety and effectiveness of the IDEAL IMPLANT in women who are undergoing primary breast augmentation or replacement of existing saline-filled or silicone gel-filled augmentation implants. | 2 mo, 6 mo, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 yrs.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Beverly Hills, California
  - Folsom, California
  - Huntington Beach, California
  - Modesto, California
  - Riverside, California
  - Sacramento, California
  - Santa Monica, California
  - Stockton, California
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Loxahatchee Groves, Florida
  - Miami, Florida
  - Ponte Vedra Beach, Florida
  - Duluth, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Allen, Texas
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - Southlake, Texas

REFERENCES:
- [Derived] Nichter LS, Hardesty RA, Anigian GM. IDEAL IMPLANT Structured Breast Implants: Core Study Results at 6 Years. Plast Reconstr Surg. 2018 Jul;142(1):66-75. doi: 10.1097/PRS.0000000000004460. PMID 29489559
- See also: Click here for more information about study: "Core Study of the Safety and Effectiveness of IDEAL IMPLANT(R) Saline-filled Breast Implants — http://www.idealimplant.com